CLINICAL TRIAL: NCT00606879
Title: A Phase I, Multi-Center, Open Label, Dose Escalation, Safety, PK and PkD Study of Orally Administered SGX523, a Small Molecule Anti-Cancer Agent, on a Twice Daily, Uninterrupted Schedule in Patients With Advanced Cancer
Brief Title: Safety Study of SGX523, a Small Molecule Met Inhibitor, to Treat Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: SGX Pharmaceuticals, Inc. (Industry)
Responsible Party: Terry Rugg, MD, SGX Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGX523-1A-002
Record Dates: First submitted 2008-01-18; First posted 2008-02-05 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Advanced Cancer
Keywords: Solid tumor; Advanced Cancer; MET inhibitor; Receptor Tyrosine Kinase Inhibitor (RTKI)
MeSH Terms: interventions — 6-(6-(1-methyl-1H-pyrazol-4-yl)-(1,2,4)triazolo(4,3-b)pyridazin-3-ylsulfanyl)quinoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: SGX523 Capsules

INTERVENTIONS:
Drug: SGX523 Capsules — This is a dose escalation study

SUMMARY:
SGX523 is a drug which acts by blocking the function of an enzyme called MET. MET activity may be important in growth and survival of some types of cancer. This Phase I trial is studying the safety, side effects, and best dose of SGX523 when given to patients with advanced cancer, and how well it inhibits MET activity in tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the ability to understand, able, willing to comply with study procedures and follow up visits, and has provided written consent
* Pathologic evidence of solid tumor
* Failed standard therapy and deemed by the Investigator to be suitable for participation into the trial
* Laboratory values (obtained within 10 days prior to enrollment): ANC: >= 1.5 × 109/L; Platelets: >= 100 × 109/L; Hemoglobin: >= 10.0 g/dL (without transfusions); Bilirubin: within normal range; AST, ALT, and alkaline phosphatase: <= 2.5 x ULN without tumor liver involvement; Serum creatinine: within normal limits; Calculated creatinine clearance: >= 60 mL/min/1.73 m2 for patients with creatinine > Institutional Normal Values; PT/PTT/INR: within normal limits..
* Have IHC evidence of phospho-MET expression on tumor material no more than 12 months old. This is a requirement only for entry into the MTD dose expansion phase.
* Have no residual toxic effects of previous therapy, and undergo a washout period of at least 5 half-lives from the time of administration of the previous therapy.

Exclusion Criteria:

* Pregnant, lactating, or may become pregnant
* Cardiac disease requiring medical therapy
* Have had a major surgery within 4 weeks prior to Day 1 of the study
* Have an active, uncontrolled bacterial, viral, or fungal infection that requires ongoing systemic therapy
* Have a known active infection with HIV, hepatitis B or C
* Have psychiatric or seizure disorders that would require therapy or interfere with study participation
* Have other severe concurrent nonmalignant disease that could compromise protocol objectives, including malabsorptive conditions
* Patients receiving prohibited medications as listed in Appendix E, including drugs categorized as strong inhibitors of CYP3A4 and A5 and drugs known to have a high potential risk of liver toxicity
* Have known allergy to SGX523 formulation or its excipients (croscarmellose sodium, lactose monohydrate and magnesium steareate)
* Patients receiving anti-coagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Within first 28 Days

SECONDARY OUTCOMES:
PK parameters: Cmin, Cmax, AUC∞, AUCtau, T1/2, Tmax, Vd, CLpo | To 28 Days after patient withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Lee Rosen, MD, Principal Investigator — Premier Onocology, California; Howard Burris, MD, Principal Investigator — Sarch Cannon Research Institute
Locations (2):
- United States (2):
  - Premier Onocology, California, Santa Monica, California
  - Sarah Cannon Research Institute, Nashville, Tennessee